CLINICAL TRIAL: NCT06659510
Title: The Effect of Transtheoretical Model-Based Education on Uncontrolled Internet Use in High School Students With Internet Addiction (Randomized Study)
Brief Title: The Effect of Transtheoretical Model-Based Education on Uncontrolled Internet Use With Internet Addiction
Acronym: internet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0000-0002-6567-9726
Record Dates: First submitted 2024-09-20; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Internet Addiction
Keywords: internet; internet addiction; uncontrolled internet use; adolescent
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Transtheoretical Mode Transtheoretical Model in Behavior Change TTM is an integrative behavior change model developed by Prochaska and Diclemente (1982). The model explains how an individual changes an unhealthy behavior or acquires a healthy behavior (Velicer et al., 2000).
  The key concept in the model is the stages of change. For this reason, the model is also called the Stages of Change Model (Marcus and Forsyth, 2009).
  This model, which allows evaluating the individual's level of readiness for change and level of self-efficacy, provides health professionals with a consultative approach that assumes that individuals have different counseling needs at different stages (Adams Fryatt, 2010).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Experimental:
  Before intervention, both Control and Face-to-face interviews were held with the intervention groups and a survey was conducted.
  and 'Descriptive questionnaire' and 'Transtheoretical Model Scale' and Young Internet Addiction Test-Short Form (YİBT-SF) Scale' were used to collect data.
  This training, conducted by the researcher, It was supported with presentations, slide shows, questions and answers, brochures and posters.
  After the training, the Intervention group After the 10-week training, they were subjected to 3-month monitoring and the follow-up process was asked at least twice a month via a social media application or by calling.
  Interventions: Other: education
- Control Group (No Intervention): As for the control group, a survey was administered via face-to-face interview method in the pre-test and post-test, but no training was given.
  In the survey application, the Diagnostic Form, Transtheoretical Model Scale and Young Internet Addiction Test Short Form Scale consist of the same questions as the survey application in the experimental group. The study continued with 38 students in the control group, as in the experimental group.

INTERVENTIONS:
Other: education — ACCORDING TO THE RESULTS AFTER THE SURVEY APPLICATION, TRAINING WAS PROVIDED TO THE ADDICTIVE STUDENTS IN THE EXPERIMENT GROUP AND MESSAGES WERE SENT FROM WHATSAPP APPLICATION IN THE FOLLOWING 2 MONTHS AFTER THE TRAINING.
  Other Names: survey application
  Arms: experimental group

SUMMARY:
Population and Sample of the Research: The population of the research consists of students who continue their education in two high schools on the Anatolian Side of Istanbul in the 2023-2024 academic year; It consists of a total of 3484 students, 742 of whom are in the 9th grade, 1173 in the 10th grade, 549 in the 11 th grade and 1020 in the 12 th grade. Stratified sampling method was used in the sampling calculation, 8 students from 9 th grades, 12 students from 10 th grades, 6 students from 11 th grades, 10 students from 12 th grades were selected, the experimental and control groups consisted of 36 students and the total sample size of the research was 72 students. has been seen.

Purpose of the Research: This study aims to examine the effect of health education based on the transtheoretical model on preventing uncontrolled internet use of high school students.

Hypotheses of the Research:

H1. The education given according to TTM provides progress in students' controlled internet usage behaviors.

H2. Education given according to TTM increases the average self-efficacy score in students.

H3. Education given according to TTM increases students' decision-making score averages.

H4. The posttest mean scores of the decision-making scale for high school students in the intervention group will be different from the control group.

H5 Post-test scores of the behavior change process scale of students in the initiative group will be different from the pre-test.

H6 There will be a difference between the self-efficacy scale mean scores of the intervention group and the scores of the control group.

DETAILED DESCRIPTION:
Type of Research: It was conducted as a pre test post test randomized controlled study to determine the effect of Transtheoretic Model Based education on high school students gaining controlled internet behavior.

Data Collection Tools:

The data of the research were collected with the Descriptive Information Form , Transtheoretic Model Scale and Young Internet Addiction Test-Short Form (YİBT-SF) Scale .

Location and Characteristics of the Research: The research will be conducted with students between the ages of 14-18 studying in two different high schools on the Anatolian Side of Istanbul. After institutional approval was obtained from the ethics committee, permission was obtained from the Provincial Directorate of National Education to conduct the study in the schools where it would be conducted. Written permission was obtained from the students and their families to conduct the research.

Type of Research: It will be carried out as a pre-test-post-test randomized controlled study in order to determine the effect of Transtheoretical Model-Based education on high school students gaining controlled internet behavior.

Population and Sample of the Research: The population of the research will be among 1749 high school students between the ages of 14-18 studying in two high schools on the Anatolian Side of Istanbul.

Accordingly, the sample of the research was determined by applying Power Analysis with the G-Power 3.1 program. According to the power analysis findings, it was determined that each group within the analysis should consist of a minimum of 30 people, with 80% power at a 95% confidence interval (or 5% significance level).

Taking into account data losses that may occur during the research process, this number was increased by 10% and as a result, it was decided that each group should consist of a minimum of 36 people. The research sample group will consist of 72 high school students between the ages of 14-18 studying in two high schools and who agree to participate in the study and meet the inclusion criteria, including 36 intervention groups and 36 control groups.

Collection of Data:

Data will be collected from individuals studying at Sarıgazi Anatolian High School and Çekmeköy Mehmetçik Anatolian High School through face-to-face interviews. Before data is collected, voluntary consents will be obtained after the necessary explanations are made to the intervention and control groups.

Data will be collected twice, as pre-test and post-test, in the intervention and control groups. The pre-test of the research was conducted between 11.09.2023-26.09.2023 and the final test was conducted between 15.03.2024-31.05.2024. The introductory information form was not applied in the post-test because the variables to be applied in the pre-test were fixed. The initiative group was provided with health training based on the stages of change model. The application lasted 6 months (3 weeks) in total.

The "Educational Program", shaped according to the "Transtheoretic Model", was carried out by face-to-face meetings with students at school. An educational program (10 weeks) and follow-up (3 months) were prepared for the students in the intervention group according to the stages of change they were in, in order to increase their level of change (decision-making and self-efficacy). No educational intervention was applied to the control group. In addition, in order to increase the effectiveness of the education, a brochure prepared specifically for each of the stages of change on "controlled internet use", formatted according to TTM, was given to the students in the intervention group immediately after the training appropriate to the stage they were in.

Implementation of the education structured according to the Transtheoretic Model. During the research process, the duration, number, content and intensity of the education given to the students in the intervention group will be determined according to the stage they are in. Students in the pre-contemplation stage will be trained at least five times, those in the contemplation stage at least four times, those in the preparation stage at least three times, those in the action stage at least twice, and those in the maintenance stage at least once. The ten-week training intervention will be delivered bi-weekly with recurring school visits, with each training lasting an average of 30-45 minutes. The final test will be administered three months after the training is completed. Training content will be prepared by researchers. The training content will include targets and approaches prepared in accordance with the stages of change. In order to determine the behavioral changes of the students in the entry group after their training is completed, students in the entry group will be called 3 times a month for 3 months (December-February), their questions will be answered and they will be motivated to take action. Students will be asked about their controlled internet use. Interviews will last approximately 10-15 minutes.

Analysis of Data:

Data will be collected in a computer environment with a statistical package program. Descriptive (percentage, ratio, arithmetic mean, standard deviation, minimum-maximum) tests and comparative analyzes will be used to evaluate the socio-demographic characteristics and scale scores of high school students in the intervention and control groups. Parametric tests will be used to ensure that the data conforms to normal distribution. One-way analysis of variance will be used in independent groups to analyze the pre-test scores of the scale and subscales of the intervention and control groups. Two-way analysis of variance will be used for repeated measurements. In the study, all results will be evaluated at a significance level of p<0.05 with a 95% confidence interval.

INITIATIVES: (Health Education with Stages of Change Model)

Stage: One of the high schools will be selected by lottery to the intervention group and the other to be the control group. Data will be collected by face-to-face interviews with students. Half of the randomly selected students will be placed in the intervention group and half in the control group. As a result of the literature review, high school students in the training initiative group, which will be created in line with the "Stages of Change Model-Based Controlled Internet Use Training Guide", will be given face-to-face training based on this guide. The training guide will be created under the following main headings in line with the Stages of Change Model:

Phase of Change (Temporal Dimension Related to Time) Change Process (Argument Dimension) Self-efficacy/Promoting Factors/Decision Making Scales (Levels of Change)

1. Change Phase (Temporary Dimension Related to Time):

   He argues that behavioral change occurs through certain stages. These stages; 1.Not thinking, 2.Contemplation, 3.Preparation, 4.Action and 5.Continuation. In the non-contemplation stage, the individual has no intention of changing his behavior in the next six months. He is not aware of the harm of his behavior. In the contemplation stage, the individual considers changing his behavior in the next six months. The positive and negative aspects of changing behavior are considered. However, the negative aspects outweigh. In the preparation phase, it intends to take action within the next month. At this stage, helmet, cycling glasses, etc. Preparations are made for change such as purchasing. In the action phase, behavioral change has occurred. Since six months have not passed since the change, there may be feedback. The maintenance phase covers the period six months after the behavioral change occurs.
2. Change Process (Independent Variable Dimension): It shows which processes (actions, behaviors, etc.) are used to progress through the stages of change. It is divided into two: cognitive and behavioral processes. While cognitive processes are used more in the non-thinking and thinking stages, behavioral processes are used more frequently in the later stages.

   cognitive processes 2.1.Awareness: It includes increasing consciousness and awareness about behavior. Trainings, conferences, comments, book reading, media and feedback methods can be used to raise awareness.

   2.2.Specific relief: It is the formation of positive emotion when the desired behavior is exhibited and negative emotion when the undesirable behavior is exhibited. Methods such as psychodrama and role playing can be used to develop this.

   2.3.Re-evaluating the environment: The impact of the behavior on the environment is evaluated cognitively and affectively. Observation can be used for this.

   2.4.Self-reevaluation: It is the process in which the individual evaluates himself. For this purpose, confrontation and interpretation techniques can be used.

   2.5.Social liberation (Environmental opportunities): Being aware of opportunities and alternatives for behavioral change enables the individual to become free and make his life easier. This includes defending rights and developing appropriate policies that support improving behavior.

   Behavioral Processes 2.1.1. Control of Stimuli (Restructuring): It includes actions that increase stimuli to initiate healthy behavior and reduce the risk of returning to undesirable behavior.

   2.2.2.Reinforcement (Reinforcing Coping/Rewarding Management): It is the use of positive reinforcers that will increase the self-efficacy of the individual by the individual himself, his friend, teacher, parent, school nurse in order to reinforce and maintain the behavioral change. For this purpose, punishment and reward methods can be applied.

   2.3.3. Agreement with Oneself (Individual Liberation / Self-Liberation): It is the process in which the individual reconsiders his decisions. Having alternatives increases the chance of success in behavioral change by giving the person freedom.

   2.4.4.Supportive Relationships (Helping Relationships): It shows the presence of those who give confidence and support for the desired behavioral change. Supporting the person in this process from family or friends is within the scope of helping relationships.

   2.5.5.Counterconditioning (Replacement): It involves learning healthy behaviors that are opposite to undesirable behavior. Behaviors that can be replaced are within the scope of counter conditioning.
3. Levels of Change Self-efficacy: It shows the individual's judgment or belief about himself/herself that he/she can perform a certain behavior successfully. It is an effective variable in starting or stopping a behavior. It is effective in the stages of the individual taking action and continuing. High self-efficacy reflects the power to stop reverting to behavior despite the pressure of incentive situations. For example; The statement "I believe that I will not eat while cycling even if I am hungry" shows that he has self-determination.

Decision Making: It reveals the perception of benefits and harms of changing behavior. The higher the perception of benefit of the individual, the more likely it is to make and maintain decisions about changing behavior. Positive aspects or The negative aspects reveal the perception of harm. For the individual in the non-thinking stage, the harms of change outweigh the benefits. For example, "When I use a reflector, I can be noticed more easily from the outside." sentence can be given as an example of decision-making based on benefit perception. (27) Phase II: Stages of Change After the Model-Based Health Education, a post-test will be administered to high school students 3 months later.

ELIGIBILITY:
Inclusion Criteria:

- Being between the ages of 14 and 18,

* Not having any mental or physical problems that would prevent participation in the study,
* No communication barriers,
* Being a student at the school where the research is conducted and obtaining voluntary consent form from the family.

Exclusion Criteria:

* Filling out the survey form incompletely.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
The analysis of the study is over | at the end of six months
  High school students with uncontrolled internet use and internet addiction were evaluated. Data were collected in the pre-test and post-test with the descriptive questionnaire (34 questions), Transtheoretical Model Scale (evaluated between 1-4 points, high scores from positive factors and perception of benefits indicate controlled internet use) and Young Internet Addiction Test Short Form (12 questions, scored between 1-5, high scores indicate addiction). Power analysis was used in the sample calculation (α=0.05, test power: 0.90, effect size: 0.76). All results in the study were at a 95% confidence interval at a significance level of p<0.05. Statistical Package for Social Sciences (SPSS) v27 and Microsoft Excel 2016 were used in the analysis of the collected data. Chi square, paired samples t, independent samples t test and Pearson correlation analysis were used in the study.
benefit of working | at the end of six months
  In the pre-test and post-test of the study, a descriptive questionnaire, the Transtheoretical Model Scale and the Young Internet Addiction Test Scale were used. Of the 76 students whose Young Internet Addiction score at the beginning of the study was 27 and above, between the ages of 14-18 and who agreed to participate in the study, 38 students were included in the experimental group and 38 students in the control group. The total follow-up lasted 6 months for each student, with 12 weeks of training and 3 months of follow-up for the 38 experimental group students. The control group was not given training and was followed up.
Benefits for students | at the end of six months
  In high school students with uncontrolled internet use and internet addiction, internet use has become controlled and addiction levels have decreased and been brought under control as a result of the study. Self-control, awareness, and individual responsibility have developed in the student. He has participated in social activities and has started to exhibit positive behaviors for his physical health (such as walking, not postponing regular nutritional needs). There has been progress in his behaviors. The student who did not think of using the internet in a controlled manner has progressed to the stages of thinking, preparing, acting, and continuing after the Controlled Internet Use training.

CONTACTS AND LOCATIONS:
Overall Officials: ARZU ŞAHİN, MASTER, Study Director — LABOR RESPONSIBLE
Locations (1):
- Marmara Üniveristesi, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The results of the study are planned to be published in an international journal and only the article and the results will be made available to other researchers, but the data will not be shared directly.

REFERENCES:
- See also: Internet addiction — https://www.who.int/news-room/questions-and-answers/item/addictive-behaviours-gaming-disorder
- See also: Addictive behaviours: Gaming disorder — https://www.who.int/news-room/questions-and-answers/item/addictive-behaviours-gaming-disorder